CLINICAL TRIAL: NCT03779698
Title: BiodentineTM Versus Formocresol Pulpotomy Technique in Primary Molars: A 12-Month Randomized Controlled Clinical Trial
Brief Title: BiodentineTM Versus Formocresol Pulpotomy Technique in Primary Molars
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Najlaa Alamoudi, Professor in Pediatric Dentistry Department, Medical Director, KAU-DH Program Director, Post Grad Studies for Master and PhD programs Program Director,of Saudi Commission for Health Specialities, Faculty of Dentistry- King Abdulaziz University, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FacultyofDentistry
Record Dates: First submitted 2018-12-13; First posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Dental Caries; Pulpotomy
Keywords: BiodentineTM; Formocresol; Primary molars; Pulpotomy
MeSH Terms: conditions — Dental Caries | interventions — formocresol

STUDY DESIGN:
Intervention Model Description: A double-blinded, split-mouth, randomized, controlled clinical study design was used with a sample of 37 healthy children aged 4- to 8-year-old. A total of 56 pairs (112 teeth) of carious primary teeth, 1 pair per child, were selected for treatment. One tooth from each pair was randomly assigned to either the BiodentineTM pulpotomy group or the formocresol pulpotomy group.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Two full-time pediatric dentistry faculty members (other than the operator) from KAU blindly evaluated all the teeth clinically and radiographically.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- BiodentineTM pulpotomy group (Experimental): A Bioactive Dentine Substitute (BiodentineTM, Septodont Ltd., Saint Maur des Faussés, France) was used following the manufacturer's recommendations. The whole pulp chamber was entirely filled with BiodentineTM until the occlusal surface.
  Interventions: Other: BiodentineTM; Drug: Formocresol
- Formocresol pulpotomy group (Active Comparator): A sterile cotton pellet moistened with 1:5 concentration formocresol (Buckley's Formocresol, Sultan Healthcare, Englewood, NJ, USA) then blotted to remove excess was placed for 5 minutes on the pulp stumps and then the pulps were covered with zinc oxide-eugenol (IRM; Dentsply, Milford, DE) dressing.
  Interventions: Other: BiodentineTM; Drug: Formocresol

INTERVENTIONS:
Other: BiodentineTM — In the experimental group, BiodentineTM was used following the manufacturer's recommendations. The whole pulp chamber was entirely filled with BiodentineTM until the occlusal surface. Follow-up was done for all children clinically at 3, 6 and 12 months and radiographically at 6 and 12 months.
  Other Names: Bioactive dentine substitute
Drug: Formocresol — In control group, a sterile cotton pellet moistened with 1:5 concentration formocresol then blotted to remove excess was placed for 5 minutes on the pulp stumps and then the pulps were covered with zinc oxide-eugenol (IRM; Dentsply, Milford, DE) dressing. Follow-up was done for all children clinically at 3, 6 and 12 months and radiographically at 6 and 12 months.
  Other Names: Buckley's Formocresol

SUMMARY:
The objective of this clinical study was to prospectively compare the clinical and radiographic success rates of BiodentineTM pulpotomies versus formocresol pulpotomies in children vital primary molars.

A randomized, split-mouth study design was used with a sample of 37 healthy children aged 4- to 8-year-old. A total of 56 pairs (112 teeth) of carious primary teeth, 1 pair per child, were selected for treatment. One tooth from each pair was randomly assigned to either the BiodentineTM pulpotomy group or the formocresol pulpotomy group. Children were followed-up at 3, 6 and 12 months for clinical evaluation and at 6 and 12 months for radiographic evaluation. Data were collected, tabulated and analyzed using Fisher exact and McNemar tests. The level of significance was set at P < 0.05.

DETAILED DESCRIPTION:
Methods This study was written according to the Consolidated Standards of Reporting Trials (CONSORT) statement.

Study design A double-blinded, split-mouth, randomized, controlled clinical study was done. Patients This study was carried out on healthy children aged 4- to 8-year-old. The children were selected from the Pediatric Dentistry Clinics, Faculty of Dentistry, King Abdulaziz University (KAU), Jeddah. Each patient had at least 2 matched bilateral carious primary molars requiring pulpotomy. Each parent signed an informed consent for the child's participation in the study. No children were excluded based on gender, race, social or economic status.

Teeth were selected based upon clinical and radiographic criteria. Teeth were unselected if any of the inclusion criteria were not met.

Preoperative periapical radiographs of the molars considered for treatment were taken using the XCP extension cone paralleling technique.

Sample size and power determination Sample size calculation for binary outcome equivalence trials was calculated using sample size calculators of a sealed envelope, randomization and online databases for clinical trials at https://www.sealedenvelope.com/power/binary-equivalence/ Thus, if there is truly no difference between the standard and experimental materials, then 102 teeth (51 for each study material) are required to be 95% sure that the limits of a two-sided 90% confidence interval will exclude a difference between the standard and experimental group of more than 10%. It is usually prudent to plan to include more than the minimum number of teeth in a study to compensate for loss during follow-up or other causes of attrition. The percentage of teeth that could be lost to follow up at all stages was set at 10% thereby forcing an increase of 5 pairs to the calculated sample size. Thus, the final sample size for this study was calculated to be 112 teeth.

Randomization Since the teeth indicated for pulpotomy must be treated as soon as possible, the patients were included at the time of diagnosis (identification) and randomization for the materials on the sides was done. In order to overcome the variable of the side preferred by the operator, the investigators made sure that both materials equally treated each side. This was performed by carrying out the block randomization technique with closed envelopes. Before recruitment of the patients, 56 sealed envelopes containing the result of randomization were prepared, sealed, and blindly mixed in a box. An envelope was for each block of two contralateral teeth (one pair). After that, the envelopes were numerated blindly from 1 to 56. The envelopes were assigned to the 56 pairs according to the beginning of the treatment (envelop number 1 was assigned to the earliest pair ready for treatment and so on). Each envelope was unsealed after the signature of the informed consent and immediately before the implementation of the first procedure on the right tooth.

One hundred and twelve molars were randomly divided into two treatment groups. Group I comprised 56 molars treated with BiodentineTM (experimental). Group II comprised 56 molars treated with formocresol (control). Each patient received 2 treatments, BiodentineTM on one side of the oral cavity and formocresol on the other side.

Procedures An operator performed the pulpotomy procedures. After application of topical anesthesia (Beutlich LP Pharmaceuticals, USA), local anesthesia was administrated using 27-gauge short needles and syringes loaded with carpules, each one contained 1.8 ml of Lidocaine 2% with epinephrine concentration of 1:100000 (Octocaine® 100, Novocol Healthcare Inc. Cambridge, Ontario, Canada). Complete isolation was performed using a rubber dam and saliva ejector. Removal of caries and deroofing of the pulp chamber were performed using a no. 330 high-speed carbide bur with copious water spray. A sharp sterile spoon excavator or a slow-speed round carbide bur (no. 6 or no. 8) was used for coronal pulp amputation. Then the pulp chamber was washed with normal saline and bleeding was controlled by placing a cotton pellet moistened with water in the pulp chamber for 5 minutes.

In the experimental group (group I), BiodentineTM (Septodont Ltd., Saint Maur des Faussés, France) was used following the manufacturer's recommendations. The whole pulp chamber was entirely filled with BiodentineTM until the occlusal surface. In control (group II), a sterile cotton pellet moistened with 1:5 concentration formocresol (Buckley's Formocresol, Sultan Healthcare, Englewood, NJ, USA) then blotted to remove excess was placed for 5 minutes on the pulp stumps and then the pulps were covered with zinc oxide-eugenol (IRM; Dentsply, Milford, DE) dressing. In both groups, all teeth were finally restored using a stainless steel crown (SSC) (3M/ESPE, St. Paul, Minn., USA).

Follow-up was done for all children clinically at 3, 6 and 12 months and radiographically at 6 and 12 months. Two full-time pediatric dentistry faculty members (other than the operator) from KAU blindly evaluated all the teeth clinically and radiographically.

Outcome assessment criteria The pulpotomy procedure was decided a clinical success if the tooth fulfilled the following criteria: (1) No pain, (2) No swelling, (3) No tenderness to percussion, (4) No abscess or fistula, and (5) No abnormal tooth mobility. The pulpotomized tooth was judged to be radiographically successful if it demonstrated the following criteria: (1) Normal periodontal ligament space (2) No periapical and furcation pathosis, and (3) No internal resorption. If pulp canal obliteration (PCO) happened, it was recorded but not considered as a treatment failure.

Statistical analysis Data were statistically analyzed using the Statistical Package for Social Sciences (SPSS) version 20.0 (SPSS Inc., Chicago, IL). Inter- and intra-examiner agreement was performed using the Kappa statistic. Fisher exact test was used to assess differences in success rates between both groups at 3, 6 or 12 months. McNemar's test was used to compare these rates in each group between pairs of follow up periods. The level of significance was set at P < 0.05.

Ethical Considerations Ethical approval was obtained from the Research Ethics Committee, Faculty of Dentistry, KAU, Jeddah, Kingdom of Saudi Arabia (Approval no. 029-14).

ELIGIBILITY:
Patient inclusion criteria:

* Patients with at least two matched bilateral deep carious primary molars indicated for pulpotomy.
* Patients within the age group of four to eight years.
* Healthy patients (both physically and mentally) without any known medical history of systemic conditions contraindicating pulp treatment.
* Cooperative patients who had behavioral ratings "positive" or "definitely positive" according to the Frankl behavior classification scale.
* Written consent was obtained from the parent/guardian after explaining the full details of the treatment procedure and its possible outcomes, discomforts, risks, and benefits.
* No patients were excluded on the basis of gender, race, social or economic background.

Patients not satisfying any of the above-mentioned criteria were excluded from the study.

Teeth inclusion criteria:

Teeth were selected based upon the following clinical and radiographic criteria: Clinically, the study included teeth with restorable crowns, teeth with pathologic carious or mechanical exposure of vital pulps and teeth with no clinical symptoms or evidence of pulp degeneration, such as spontaneous or nocturnal pain, pain on percussion, history of swelling, or sinus tracts and teeth with no tenderness to percussion, physiologic or pathologic mobility. Radiographically, the recruited teeth should have a normal radiographic appearance with healthy supporting tissues, no signs of internal resorption, or pathologic external root resorption and no periapical or inter-radicular pathosis, with at least two-thirds of the root remaining (not more than one-third of the root is physiologically resorbed).

Teeth exclusion criteria:

Teeth were excluded if (1) any of the above-mentioned clinical or radiographic inclusion criteria were not satisfied, (2) hemostasis could not be achieved within 5 minutes by direct contact with a wet cotton pellet, prior to material placement, or (3) the remaining radicular tissue was non-vital (with suppuration or purulence necrosis).

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Clinical evaluation of BiodentineTM and formocresol pulpotomies 3 months after treatment | After 3 months
  Clinical evaluation of BiodentineTM and formocresol pulpotomies was performed 3 months after treatment using the preset clinical criteria. The pulpotomy procedure was decided a clinical success if the tooth fulfilled the following criteria: (1) No pain, (2) No swelling, (3) No tenderness to percussion, (4) No abscess or fistula, and (5) No abnormal tooth mobility.
Clinical evaluation of BiodentineTM and formocresol pulpotomies 6 months after treatment | After 6 months
  Clinical evaluation of BiodentineTM and formocresol pulpotomies was performed 6 months after treatment using the preset clinical criteria. The pulpotomy procedure was decided a clinical success if the tooth fulfilled the following criteria: (1) No pain, (2) No swelling, (3) No tenderness to percussion, (4) No abscess or fistula, and (5) No abnormal tooth mobility.
Clinical evaluation of BiodentineTM and formocresol pulpotomies 12 months after treatment | After12 months
  Clinical evaluation of BiodentineTM and formocresol pulpotomies was performed 12 months after treatment using the preset clinical criteria. The pulpotomy procedure was decided a clinical success if the tooth fulfilled the following criteria: (1) No pain, (2) No swelling, (3) No tenderness to percussion, (4) No abscess or fistula, and (5) No abnormal tooth mobility.
Radiographic evaluation of BiodentineTM and formocresol pulpotomies 6 months after treatment | After 6 months
  Radiographic evaluation of BiodentineTM and formocresol pulpotomies was performed 6 months after treatment using periapical radiographs. The pulpotomized tooth was judged to be radiographically successful if it demonstrated the following criteria: (1) Normal periodontal ligament space (2) No periapical and furcation pathosis, and (3) No internal resorption. If pulp canal obliteration (PCO) happened, it was recorded but not considered as a treatment failure.
Radiographic evaluation of BiodentineTM and formocresol pulpotomies 12 months after treatment | After 12 months
  Radiographic evaluation of BiodentineTM and formocresol pulpotomies was performed 12 months after treatment using periapical radiographs. The pulpotomized tooth was judged to be radiographically successful if it demonstrated the following criteria: (1) Normal periodontal ligament space (2) No periapical and furcation pathosis, and (3) No internal resorption. If pulp canal obliteration (PCO) happened, it was recorded but not considered as a treatment failure.

CONTACTS AND LOCATIONS:
Overall Officials: Najlaa M Alamoudi, BDS,MSc,DSc, Principal Investigator — King Abdulaziz University, Faculty of Dentistry
Locations (1):
- King Abdulaziz University, Faculty of Dentistry, Jeddah, Mecca Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Erdem AP, Guven Y, Balli B, Ilhan B, Sepet E, Ulukapi I, Aktoren O. Success rates of mineral trioxide aggregate, ferric sulfate, and formocresol pulpotomies: a 24-month study. Pediatr Dent. 2011 Mar-Apr;33(2):165-70. PMID 21703067
- [Background] Agamy HA, Bakry NS, Mounir MM, Avery DR. Comparison of mineral trioxide aggregate and formocresol as pulp-capping agents in pulpotomized primary teeth. Pediatr Dent. 2004 Jul-Aug;26(4):302-9. PMID 15344622
- [Background] Farsi N, Alamoudi N, Balto K, Mushayt A. Success of mineral trioxide aggregate in pulpotomized primary molars. J Clin Pediatr Dent. 2005 Summer;29(4):307-11. doi: 10.17796/jcpd.29.4.n80t77w625118k73. PMID 16161395
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. Int J Surg. 2011;9(8):672-7. doi: 10.1016/j.ijsu.2011.09.004. Epub 2011 Oct 13. No abstract available. PMID 22019563
- [Background] Sonmez D, Sari S, Cetinbas T. A Comparison of four pulpotomy techniques in primary molars: a long-term follow-up. J Endod. 2008 Aug;34(8):950-5. doi: 10.1016/j.joen.2008.05.009. PMID 18634926
- [Background] Fuks AB, Bimstein E, Guelmann M, Klein H. Assessment of a 2 percent buffered glutaraldehyde solution in pulpotomized primary teeth of schoolchildren. ASDC J Dent Child. 1990 Sep-Oct;57(5):371-5. PMID 2120303
- [Derived] El Meligy OAES, Alamoudi NM, Allazzam SM, El-Housseiny AAM. BiodentineTM versus formocresol pulpotomy technique in primary molars: a 12-month randomized controlled clinical trial. BMC Oral Health. 2019 Jan 7;19(1):3. doi: 10.1186/s12903-018-0702-4. PMID 30612569